CLINICAL TRIAL: NCT02195700
Title: A Randomized, Double-Blind, Placebo-Controlled Study of SD-809 (Deutetrabenazine) for the Treatment of Moderate to Severe Tardive Dyskinesia
Brief Title: Aim to Reduce Movements in Tardive Dyskinesia
Acronym: ARM-TD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Auspex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SD-809-C-18
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Tardive Dyskinesia
Keywords: Dyskinesias; Movement Disorders; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations; Signs and Symptoms
MeSH Terms: conditions — Tardive Dyskinesia; Dyskinesias; Movement Disorders; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations; Signs and Symptoms | interventions — deutetrabenazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SD-809 (Experimental): SD-809 tablets taken twice daily for 12 weeks.
  Interventions: Drug: SD-809
- Sugar Pill (Placebo Comparator): Placebo tablets taken twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SD-809 — SD-809 tablets taken twice daily for 12 weeks, includes a dose titration period and maintenance period.
  Other Names: deutetrabenazine; AUSTEDO®
  Arms: SD-809
Drug: Placebo — Placebo tablets taken twice daily for 12 weeks.
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to determine whether an investigational drug, SD-809 (deutetrabenazine), will reduce the severity of abnormal involuntary movements of tardive dyskinesia.

ELIGIBILITY:
Inclusion Criteria:

* History of using a dopamine receptor antagonist for at least 3 months
* Clinical diagnosis of tardive dyskinesia and has had symptoms for at least 3 months prior to screening
* Subjects with underlying psychiatric diagnosis are stable and have no change in psychoactive medications
* Have a mental health provider and does not anticipate any changes to treatment regimen in the next 3 months
* History of being compliant with prescribed medications
* Able to swallow study drug whole
* Be in good general health and is expected to attend all study visits and complete study assessments
* Female subjects must not be pregnant and agree to an acceptable method of contraception

Exclusion Criteria:

* Currently receiving medication for the treatment of tardive dyskinesia
* Have a neurological condition other than tardive dyskinesia that may interfere with assessing the severity of dyskinesias
* Have a serious untreated or undertreated psychiatric illness
* Have recent history or presence of violent behavior
* Have unstable or serious medical illness
* Have evidence of hepatic impairment
* Have evidence of renal impairment
* Have known allergy to any component of SD-809 or tetrabenazine
* Has participated in an investigational drug or device trial and received study drug within 30 days
* Have acknowledged use of illicit drugs
* Have a history of alcohol or substance abuse in the previous 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, M.D., Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (41):
- United States (32):
  - Tuscaloosa, Alabama
  - Anaheim, California
  - Glendale, California
  - Oceanside, California
  - Orange, California
  - San Bernardino, California
  - San Diego, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Gainesville, Florida
  - Lake City, Florida
  - Miami, Florida
  - Orlando, Florida
  - Port Charlotte, Florida
  - Chicago, Illinois
  - Baltimore, Maryland
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Asheville, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Fort Worth, Texas
  - Salt Lake City, Utah
- Prague, Czechia
- Poland (6):
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Torun
- Slovakia (2):
  - Domaša
  - Rožňava

REFERENCES:
- [Derived] Frank S, Anderson KE, Fernandez HH, Hauser RA, Claassen DO, Stamler D, Factor SA, Jimenez-Shahed J, Barkay H, Wilhelm A, Alexander JK, Chaijale N, Barash S, Savola JM, Gordon MF, Chen M. Safety of Deutetrabenazine for the Treatment of Tardive Dyskinesia and Chorea Associated with Huntington Disease. Neurol Ther. 2024 Jun;13(3):655-675. doi: 10.1007/s40120-024-00600-1. Epub 2024 Apr 1. PMID 38557959

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 202 patients were screened and gave informed consent to enter the study. 85 were either ineligible for entry into the study or declined study participation. The most common reason for ineligibility (49 patients) was insufficient TD severity as assessed with Abnormal Involuntary Movement Scale (AIMS). 117 patients were randomized.
Groups:
- SD-809: Patients underwent dose adjustment of SD-809 over the initial 6 weeks of treatment, starting treatment with SD-809 at 6 mg twice daily and titrating to a maximum total daily dose of 48 mg per day. The optimal dose was continued by a 6-week maintenance period, which was followed by a 1-week washout.
  Patients who completed the study had the option to rollover into a long-term safety study (Study SD-809-C-20, NCT02198794). For patients who did not enter the long-term safety study, there was an additional 3-week safety follow-up period after treatment.
- Placebo: Patients underwent 'dose adjustment' of placebo over the initial 6 weeks of treatment. The optimal dose was continued by a 6-week maintenance period, which was followed by a 1-week washout. Patients who completed the study had the option to rollover into a long-term safety study (Study SD-809-C-20, NCT02198794). For patients who did not enter the long-term safety study, there was an additional 3-week safety follow-up period after treatment.
Period: Overall Study
Arm/Group | SD-809 | Placebo
Started | 58 | 59
Safety and ITT Populations | 58 | 59
Modified ITT Population | 56 (ITT who received study drug and >=1 centrally read post-baseline AIMS from weeks 2, 4, 6, 9, or 12) | 57 (ITT who received study drug and >=1 centrally read post-baseline AIMS from weeks 2, 4, 6, 9, or 12)
Maintenance Period | 53 | 54
Completed | 52 | 52
Not Completed | 6 | 7
Not completed — Protocol Violation | 0 | 2
Not completed — Noncompliance | 1 | 0
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | SD-809 | Placebo | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.82) | 53.3 (10.64) | 54.6 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 61
  Male | 29 | 27 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 11 | 15
  Not Hispanic or Latino | 53 | 47 | 100
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 14 | 33
  White | 37 | 44 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education Level [Count of Participants; unit: Participants]
  =12 years or fewer of formal education | 30 | 30 | 60
  >12 years of formal education | 28 | 29 | 57
Weight [Mean (Standard Deviation); unit: kg] | 86.94 (24.081) | 84.95 (20.975) | 85.94 (22.493)
Height [Mean (Standard Deviation); unit: cm] | 169.23 (11.462) | 169.72 (10.098) | 169.48 (10.752)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.35 (7.926) | 29.45 (6.958) | 29.89 (7.435)
Using a Dopamine Receptor Antagonist (DRA) [Count of Participants; unit: Participants] — The randomization was stratified by baseline use of DRA (currently taking versus not currently taking a DRA).
  Participants
    Yes | 45 | 49 | 94
    No | 13 | 10 | 23
Duration of tardive dyskinesia [Mean (Standard Deviation); unit: months] | 72.6 (81.65) | 76.8 (82.05) | 74.7 (81.53)
Centrally Read Abnormal Involuntary Movement Scale (AIMS) Score [Mean (Standard Deviation); unit: units on a scale] — AIMS is an assessment tool used to detect and follow the severity of TD over time. The AIMS is composed of 12 clinician-administered and scored items. AIMS was digitally video recorded using a standard protocol and independently reviewed by blinded central raters who were experts in movement disorders.
  This data sums items 1 through 7 which cover orofacial movements, and extremity and truncal dyskinesia. Severity ratings were from 0 (none) to 4 (severe) for a total scale of 0 (no orofacial, truncal, and extremity dyskinesia) to 28 (severe orofacial, truncal, and extremity dyskinesia). Population: Central reading was not available for one placebo patient.
  units on a scale
    number analyzed (Participants) | 58 | 58 | 116
    (all) | 9.6 (4.07) | 9.6 (3.77) | 9.6 (3.90)
Modified Craniocervical Dystonia Questionnaire (CDQ-24) [Mean (Standard Deviation); unit: units on a scale] — The CDQ-24 is a disease-specific quality of life questionnaire developed for use in patients with craniocervical dystonia, including both cervical dystonia (CD) and blepharospasm (BPS). The CDQ 24 was modified such that the questions focus more directly on the impact of TD (as opposed to CD/BPS) on quality of life. Each of the 24 questions was rated by patients on a scale of 0=no impairment to 4=severest impairment for a total scale of 0 (no impairment) to 96 (severe impairment). Population: Baseline CDQ-24 was not completed by two placebo patients.
  units on a scale
    number analyzed (Participants) | 58 | 57 | 115
    (all) | 38.4 (20.41) | 39.7 (18.17) | 39.1 (19.26)

OUTCOME MEASURES:

1. Primary Outcome: Change in Centrally Read Abnormal Involuntary Movement Scale (AIMS) Score From Baseline to Week 12 Using Mixed Model Repeated Measures (MMRM) Analysis
Description: AIMS is an assessment tool used to detect and follow the severity of TD over time. The AIMS is composed of 12 clinician-administered and scored items. AIMS was digitally video recorded using a standard protocol and independently reviewed by blinded central raters who were experts in movement disorders.
  This outcome sums items 1 through 7 which cover orofacial movements, and extremity and truncal dyskinesia. Severity ratings were from 0 (none) to 4 (severe) for a total scale of 0 (no orofacial, truncal, and extremity dyskinesia) to 28 (severe orofacial, truncal, and extremity dyskinesia). A negative change from baseline score indicates improvement.
  A MMRM analysis with change from baseline in AIMS score as dependent variable was used. The model included fixed effects for treatment, time point, treatment-by-time point interaction, DRA status, and baseline AIMS as a covariate. An unstructured covariance model was used.
Time Frame: Day 0 (Baseline), Weeks 2, 4, 6, 9 and 12
Population: The Modified ITT (mITT) Population was defined as all patients in the ITT Population who received study drug and had at least 1 centrally read post-baseline assessment of the AIMS from at least 1 scheduled post-baseline time point. Number analyzed includes participants who had week 12 readings minus one placebo patient missing a baseline reading.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SD-809 | Placebo
Number analyzed (Participants) | 52 | 51
units on a scale | -3.0 (0.45) | -1.6 (0.46)
Statistical Analysis 1: Comparison: SD-809 vs Placebo; The linear mixed model for repeated measurements (MMRM) included fixed effects for treatment, each scheduled time point (5 levels: weeks 2, 4, 6, 9, and 12), the treatment-by-time point interaction, and the DRA status. Baseline AIMS score was a covariate. The unstructured covariance model was used, and the primary analysis compared the SD-809 and placebo groups at week 12. This was based on the F-test using the Satterhwaite method to compute the denominator degrees of freedom; Test type: Superiority; p = 0.0188, unstructured covariance — 5% level of significance (2-sided); LSM difference = -1.4, 95% CI 2-sided [-2.6 to -0.2], Standard Error of Mean 0.60

2. Secondary Outcome: Percentage of Patients Who Are a Treatment Success at Week 12 as Assessed by the Clinical Global Impression of Change (CGIC)
Description: The CGIC is a single-item questionnaire that asks the investigator to assess a patient's TD symptoms at specific visits after initiating therapy. The CGIC uses a 7 point Likert Scale, ranging from very much worse (-3) to very much improved (+3), to assess overall response to therapy. A treatment success was defined as "much improved" or "very much improved" at the week 12 visit. Patients whose status at week 12 was not known, as well as patients who were not "much improved" or "very much improved" at the week 12 visit, were considered treatment failures.
Time Frame: Week 12
Population: modified intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | SD-809 | Placebo
Number analyzed (Participants) | 56 | 57
percentage of participants | 48.2 | 40.4
Statistical Analysis 1: Comparison: SD-809 vs Placebo; The secondary efficacy endpoints were analyzed using a hierarchical testing procedure. If the primary analysis was statistically significant (p<0.05), then the first key secondary endpoint was to be analyzed. If the first key secondary endpoint was statistically significant, then the second key secondary endpoint was to be similarly analyzed. For any analysis that was not statistically significant, all subsequent analyses of key secondary endpoints were exploratory rather than confirmatory; Test type: Superiority; p = 0.4001, Pearson's chi-square test — 5% level of significance (2-sided); Differences in % = 7.9, 95% CI 2-sided [-10.2 to 25.2]

3. Secondary Outcome: Percentage of Patients Who Are a Treatment Success at Week 12 as Assessed by the Patient Global Impression of Change (PGIC)
Description: The PGIC is a single-item questionnaire that asks the patient to assess their TD symptoms at specific visits after initiating therapy. The PGIC uses a 7 point Likert Scale, ranging from very much worse (-3) to very much improved (+3), to assess overall response to therapy. A treatment success was defined as "much improved" or "very much improved" at the week 12 visit. Patients whose status at week 12 was not known, as well as patients who were not "much improved" or "very much improved" at the week 12 visit, were considered treatment failures.
Time Frame: Week 12
Population: modified intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | SD-809 | Placebo
Number analyzed (Participants) | 56 | 57
percentage of participants | 42.9 | 29.8

4. Secondary Outcome: Change From Baseline to Week 12 in the Modified Craniocervical Dystonia Questionnaire (CDQ-24)
Description: The CDQ-24 is a disease-specific quality of life questionnaire developed for use in patients with craniocervical dystonia, including both cervical dystonia (CD) and blepharospasm (BPS). The CDQ 24 was modified such that the questions focus more directly on the impact of TD (as opposed to CD/BPS) on quality of life. The following domains are evaluated in the CDQ-24: stigma, emotional well-being, pain, activities of daily living, and social/family life. Each of the 24 questions were rated by patients on a scale of 0=no impairment to 4=severest impairment for a total scale of 0 (no impairment) to 96 (severe impairment). Negative change from baseline scores indicate improvement.
Time Frame: Day 0 (Baseline), Week 12 with last observation carried forward
Population: modified intent to treat population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SD-809 | Placebo
Number analyzed (Participants) | 56 | 57
units on a scale | -11.1 (2.14) | -8.3 (2.31)

5. Secondary Outcome: Participants With Adverse Events for the Overall Treatment Period
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator and includes possibly, probably and definitely related categories. Serious AEs (SAE) include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | SD-809 | Placebo
Number analyzed (Participants) | 58 | 59
Participants
  Overall Treatment Period: any AE | 41 | 36
  Overall Treatment Period: SAE | 3 | 5
  Overall Treatment Period: Severe AE | 3 | 3
  Overall Treatment Period: treatment-related AE | 28 | 21
  Overall Treatment Period: Deaths | 0 | 0

6. Secondary Outcome: Percentage Change in Centrally Read Abnormal Involuntary Movement Scale (AIMS) Score From Baseline to Week 12 Using MMRM Analysis
Description: AIMS is an assessment tool used to detect and follow the severity of TD over time. The AIMS is composed of 12 clinician-administered and scored items. AIMS was digitally video recorded using a standard protocol and independently reviewed by blinded central raters who were experts in movement disorders.
  This outcome sums items 1 through 7 which cover orofacial movements, and extremity and truncal dyskinesia. Severity ratings were from 0 (none) to 4 (severe) for a total scale of 0 (no orofacial, truncal, and extremity dyskinesia) to 28 (severe orofacial, truncal, and extremity dyskinesia). A negative percent change from baseline score indicates improvement.
  The MMRM model includes fixed effects for treatment, time point (weeks 2, 4, 6, 9, 12), treatment-by-time point interaction, DRA status, and baseline AIMS as a covariate. Patient is a random effect.
Time Frame: Day 0 (Baseline), Weeks 2, 4, 6, 9 and 12
Population: modified intent to treat population. Number analyzed includes participants who had week 12 readings minus one placebo patient missing a baseline reading.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | SD-809 | Placebo
Number analyzed (Participants) | 52 | 51
percentage change | -26.7 (6.06) | -15.5 (6.26)

7. Secondary Outcome: Cumulative Percentage of Abnormal Involuntary Movement Scale (AIMS) Responders by Response Level (Percentage Improvement From Baseline) at Week 12
Description: Response level represents the % improvement in AIMS from baseline. AIMS is an assessment tool used to detect and follow the severity of TD over time. The AIMS is composed of 12 clinician-administered and scored items. AIMS was digitally video recorded using a standard protocol and independently reviewed by blinded central raters who were experts in movement disorders.
  This outcome sums items 1 through 7 which cover orofacial movements, and extremity and truncal dyskinesia. Severity ratings were from 0 (none) to 4 (severe) for a total scale of 0 (no orofacial, truncal, and extremity dyskinesia) to 28 (severe orofacial, truncal, and extremity dyskinesia).
  Patients with a missing AIMS score were considered to be AIMS nonresponders.
Time Frame: Day 0 (Baseline), Week 12
Population: modified intent to treat population.
Measure: Number; unit: percentage of participants
Arm/Group | SD-809 | Placebo
Number analyzed (Participants) | 56 | 57
percentage of participants
  >=10% | 69.6 | 42.1
  >=20% | 50.0 | 29.8
  >=30% | 46.4 | 24.6
  >=40% | 32.1 | 22.8
  >=50% | 23.2 | 17.5
  >=60% | 19.6 | 8.8
  >=70% | 10.7 | 1.8
  >=80% | 8.9 | 1.8
  >=90% | 3.6 | 1.8

8. Secondary Outcome: Change in Locally Read Abnormal Involuntary Movement Scale (AIMS) Score From Baseline to Week 12 Using MMRM Analysis
Description: This outcome is similar to the primary outcome except that AIMS was read locally.
  AIMS is an assessment tool used to detect and follow the severity of TD over time. The AIMS is composed of 12 clinician-administered and scored items. This outcome reports the local reading of AIMS data.
  This outcome sums items 1 through 7 which cover orofacial movements, and extremity and truncal dyskinesia. Severity ratings were from 0 (none) to 4 (severe) for a total scale of 0 (no orofacial, truncal, and extremity dyskinesia) to 28 (severe orofacial, truncal, and extremity dyskinesia). A negative change from baseline score indicates improvement.
  A MMRM analysis with change from baseline in AIMS score as dependent variable was used. The model included fixed effects for treatment, time point (weeks 2, 4, 6, 9, and 12), treatment-by-time point interaction, DRA status, and baseline AIMS as a covariate.
Time Frame: Day 0 (Baseline), Weeks 2, 4, 6, 9 and 12
Population: modified intent to treat analysis. Number analyzed includes participants who had week 12 readings minus one placebo patient missing a baseline reading.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SD-809 | Placebo
Number analyzed (Participants) | 52 | 51
units on a scale | -4.9 (0.64) | -3.7 (0.65)

ADVERSE EVENTS:
Time Frame: Day 1 to Week 12
Arm/Group | SD-809 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 3/58 | 5/59
Other Adverse Events (participants affected / at risk) | 24/58 | 26/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SD-809 (N=58) | Placebo (N=59)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Laryngeal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SD-809 (N=58) | Placebo (N=59)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 4 (4) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 3 (3)
Somnolence (Nervous system disorders) | 8 (8) | 6 (8)
Headache (Nervous system disorders) | 3 (3) | 6 (6)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Akathisia (Nervous system disorders) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.